CLINICAL TRIAL: NCT04961853
Title: Diagnostic Value of Hand Ultrasound Versus MRI in Rheumatoid Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fady Boles Anwer, resident doctor at Diagnostic and Interventional Radiology, Sohag university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-21-07-12
Record Dates: First submitted 2021-07-13; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Patient's With Rheumatoid Arthritis
MeSH Terms: interventions — High-Energy Shock Waves; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cases (Experimental)
  Interventions: Radiation: Ultrasound and MRI

INTERVENTIONS:
Radiation: Ultrasound and MRI — Ultrasound examination and magnetic resonance imaging on the hand

SUMMARY:
Rheumatoid arthritis (RA) is one of the most common autoimmune rheumatic diseases, affecting one in 100 individuals worldwide. It is considered a complex systemic multifactorial inflammatory process in which the immune system targets synovial joints and causes mild to severe joint destruction with extra-articular manifestations.

If left untreated, RA leads to deformity, considerable disability, and major comorbid conditions, including cardiovascular disease and increased mortality.

Early treatment with targeted therapies can alter long-term outcomes by minimizing disease activity, preventing joint damage and disability, and improving patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Adult-onset disease.
2. Patients who fulfill the 2010 American College of Rheumatology/European League Against Rheumatism classification criteria for rheumatoid arthritis.

Exclusion Criteria:

1. Any patient with any collagen disease rather than Rheumatoid arthritis.
2. Patients with joints deformities.
3. Patient's with implanted metal clips or wires or artificial pacemaker.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of Ultrasound and MRI in Rheumatoid Arthritis of the hand | 3 months
  determine the diagnostic value and associated weakness and strength aspects of hand ultrasound versus MRI in patients with rheumatoid arthritis, particularly in early disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaeley GS, Bakewell C, Deodhar A. The importance of ultrasound in identifying and differentiating patients with early inflammatory arthritis: a narrative review. Arthritis Res Ther. 2020 Jan 2;22(1):1. doi: 10.1186/s13075-019-2050-4. PMID 31898524
- [Background] Tan YK, Ostergaard M, Conaghan PG. Imaging tools in rheumatoid arthritis: ultrasound vs magnetic resonance imaging. Rheumatology (Oxford). 2012 Dec;51 Suppl 7:vii36-42. doi: 10.1093/rheumatology/kes329. PMID 23230093
- [Background] Hodgson RJ, O'Connor P, Moots R. MRI of rheumatoid arthritis image quantitation for the assessment of disease activity, progression and response to therapy. Rheumatology (Oxford). 2008 Jan;47(1):13-21. doi: 10.1093/rheumatology/kem250. Epub 2007 Nov 28. PMID 18045811
- [Background] Rowbotham EL, Grainger AJ. Rheumatoid arthritis: ultrasound versus MRI. AJR Am J Roentgenol. 2011 Sep;197(3):541-6. doi: 10.2214/ajr.11.6798. PMID 21862794